CLINICAL TRIAL: NCT04889027
Title: Turkish Validity and Reliability of Standardized Infant NeuroDevelopmental Assessment
Brief Title: Standardized Infant NeuroDevelopmental Assessment (SINDA) in 0-24 Months Age in Turkey
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Pt, PhD, Associate Professor, Ondokuz Mayıs University
Other Study IDs: 2020/017
Record Dates: First submitted 2021-05-10; First posted 2021-05-17 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Infant, Premature, Diseases; Motor Development
Keywords: infant; validty; neurologic examination; motor development
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Standardized Infant NeuroDevelopmental Assessment — The neurological scale of SINDA is designed as a screening tool as follows: (1) in the first year of life after the neonatal period, that is, in the corrected age range of 6 weeks to 12 months; (2) covers all infant neurological areas; (3) it is standardized, that is, it has a set of items and criteria identical to that age range; (4) results in a score that is largely independent of the baby's age; (5) general pediatricians are easy to use and take about 10 minutes to do (including recording scores); (6) contains a substantial part of items assessing the quality of spontaneous movements; and (7) helps predict developmental outcome (Hadder-Algra et al., 2018).
  Other Names: Alberta Infant Motor Scale (AIMS); Hammersmith Infant Neurological Examination (HINE)

SUMMARY:
This study aims to assess Turkish validity and reliability of Standardized Infant Neurodevelopmental Assessment and to spread its use for evaluation in early rehabilitation in our country.

DETAILED DESCRIPTION:
There are developments in the field of diagnosing children with a high risk of developmental disorders such as cerebral palsy (CP), mental problems and autism spectrum disorder in infancy. In particular, in infants experiencing the onset of extrauterine life in the neonatal intensive care unit, the combination of neonatal neuroimaging along with the assessment of general movements results in a highly accurate prediction of CP .

A clinical tool often used in predictions is a neurological examination. Various standard variants are available, such as the Hammersmith Infant Neurological Examination (HINE), Alberta Infant Motor Scale (AIMS).

The neurological scale of SINDA is designed as a screening tool as follows: (1) in the first year of life after the neonatal period, that is, in the corrected age range of 6 weeks to 12 months; (2) covers all infant neurological areas; (3) it is standardized, that is, it has a set of items and criteria identical to that age range; (4) results in a score that is largely independent of the baby's age; (5) general pediatricians are easy to use and take about 10 minutes to do (including recording scores); (6) contains a substantial part of items assessing the quality of spontaneous movements; and (7) helps predict developmental outcome .This study aims to assess Turkish validity and reliability of Standardized Infant Neurodevelopmental Assessment and to spread its use for evaluation in early rehabilitation in our country.

ELIGIBILITY:
Inclusion Criteria:

* at-risk infants
* discharged from neonatal intensive care unit;
* age between 0 - 24 months old (corrected age for premature infants);
* having a family acceptance for the participation

Exclusion Criteria:

* having congenital anomalies,
* musculoskeletal disorders,
* cyanotic congenital heart disease and
* mechanical dependency

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: At-risk infant between 0-24 months (adjusted age will be calculated for premature babies), who are followed as neurologically and developmentally, whose medical treatments have been completed and who are not in neonatal intensive care will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Standardized Infant NeuroDevelopmental Assessment | 20-30 minutes
  The neurological scale of SINDA is designed as a screening tool as follows: (1) in the first year of life after the neonatal period, that is, in the corrected age range of 6 weeks to 12 months; (2) covers all infant neurological areas; (3) it is standardized, that is, it has a set of items and criteria identical to that age range; (4) results in a score that is largely independent of the baby's age; (5) general pediatricians are easy to use and take about 10 minutes to do (including recording scores); (6) contains a substantial part of items assessing the quality of spontaneous movements; and (7) helps predict developmental outcome

SECONDARY OUTCOMES:
Hammersmith Infant Neurological Examination (HINE) | 30-40 minutes
  The HINE includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour. The first section evaluates cranial nerve, posture, movements, tone and reflexes. These items are not age-dependent. The second section evaluates head control, sitting, voluntary grasping, rolling, crawling and walking. The third section evaluates state of consciousness, emotional state and social orientation.
Alberta Infant Motor Scale (AIMS). | 30-45 minutes
  This scale is a norm-referenced observational tool designed for the evaluation of gross motor development in infants from birth to 18 months of age or the acquisition of independent walking. It consists of 58 items and four subscales: supine (9 items), prone (21 items), sitting (12 items) and standing (16 items), which are observed in postural alignment, antigravity movements and surface contact.

CONTACTS AND LOCATIONS:
Overall Officials: NILAY ÇÖMÜK BALCI, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Nilay Çömük Balci, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No